CLINICAL TRIAL: NCT06201832
Title: Prevalence of Cardiac Amyloidosis in Heart Failure Patients With Preserved Left Ventricular Ejection Fraction in Tunisia
Brief Title: Cardiac Amyloidosis in HFpEF Tunisian Patients
Acronym: Amy-Card
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Lilia Zakhama, Professor, University Tunis El Manar
Other Study IDs: 13-2023
Record Dates: First submitted 2023-12-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Amyloidosis; Heart Failure With Preserved Ejection Fraction; Echocardiography; CMR; Bone Scintigraphy; Prevalence; Diagnosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiac amyloidosis (CA) has recently been reported as a common cause of heart failure with preserved left ventricular ejection fraction (HFpEF), with a prevalence of 6% in elderly HFpEF patients. However, the diagnosis of CA is still challenging and requires multiple costly investigations.

Regardless of the type of CA, TTR or AL, early diagnosis significantly improves prognosis.

In this study, the investigators aimed to determine the prevalence of CA in Tunisian HFpEF patients and to identify clinical and ultrasound criteria predictive of CA.

ELIGIBILITY:
Inclusion Criteria:

* HFpEF during the previous year
* IVS thickness of 12mm or greater

Exclusion Criteria:

* age under 60 years
* Acute coronary syndrome complicated by HFpEF
* Congenital heart disease

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 60 years or older, admitted to hospital for HFpEF in the preceding year, and with an IVS thickness of 12 mm or greater.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of cardiac amyloidosis among HFpEF old Tunisian Patients | one year
  Prevalence of cardiac amyloidosis in a Tunisian cohort of HFpEF patients aged 60 years or older with interventricular septal thickness equal to or greater than 12 mm

SECONDARY OUTCOMES:
Identify imaging criteria predictive of cardiac amyloidosis on CMR and echocardiography | one year
  Number of cardiac amyloidosis patients with impaired global longitudinal left ventricular strain and/or impaired left atrial strain on echocardiography and/or elevated extra cellular volume (ECV) on CMR.
Frequency of different types of cardiac amyloidosis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Lilia Zakhama, Prof, Principal Investigator — University of Tunis El Manar, Faculty of Medicine of Tunis, Tunisia
Locations (1):
- Security Hospital Forces, La Marsa, Tunis Governorate, Tunisia